CLINICAL TRIAL: NCT03954431
Title: Study of High-resolution, Lower Dose Dedicated Breast CT.
Brief Title: High-Resolution Lower Dose Dedicated Breast Computed Tomography (CT)
Acronym: LowerDoseBCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1903399639; R01CA199044 (NIH)
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All subjects will undergo a bilateral breast CT (BCT) exam.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Dedicated breast computed tomography (BCT) (Experimental): All subjects will undergo bilateral breast CT (BCT) imaging exam.
  Interventions: Diagnostic Test: Dedicated breast CT(BCT)

INTERVENTIONS:
Diagnostic Test: Dedicated breast CT(BCT) — The breast CT device will take multiple pictures of the subject's uncompressed breast and creates a 3-D image of the breast.
  Other Names: BCT

SUMMARY:
This study is being performed to find out if a new kind of breast imaging (called dedicated breast CT or BCT) can help doctors to see the small structures in breast tissue more clearly. The investigators also want to find out if using the BCT will provide a more accurate diagnosis of breast cancer.

DETAILED DESCRIPTION:
The breast imaging device that will be used in this study (breast computed tomography or BCT) is not FDA-approved for this use so this is a research study. The machine has been redesigned to see if doctors can see smaller structures and use a lower radiation dose.

The breast CT device will take multiple pictures of the subject's breast and create a 3-D image of the breast. It does not compress or squash the breast like a mammogram.

ELIGIBILITY:
Inclusion criteria: All subjects that are eligible to participate in the study will be women who satisfy all of the inclusion criteria stated below:

* who are 40 years of age or older (typical screening age range)
* who are undergoing or scheduled for screening or diagnostic imaging, or need a biopsy to investigate an abnormality in the breast.

Exclusion criteria: Subjects that present with any of the criteria listed below will be excluded:

* Males,
* women less than 40 years old,
* women unable to self-consent,
* prisoners,
* pregnant, suspected to be pregnant, or lactating women (self-reported)
* women with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker;
* women who are unable to tolerate study constraints, frail, or unable to cooperate;
* women who weigh more than 440 lbs (200 Kg), which is the weight limit for the patient support table of the BCT system;
* women who have received radiation treatments to the thorax for malignant and nonmalignant conditions, such as (but not limited to) treatment for enlarged thymus gland as an infant, irradiation for benign breast conditions, including breast inflammation after giving birth, and treatment for Hodgkin's disease;
* women who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram;
* women who have received large number of diagnostic x-ray examinations for monitoring of disease such as (but not limited to) tuberculosis, and severe scoliosis.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 12 months after completion of accrual
  The diagnostic accuracy of BCT will be determined from a multi-reader, multi-case reader study.

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Vedantham, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States